CLINICAL TRIAL: NCT07246863
Title: Ph 2, Randomized, Blinded, Placebo-Controlled Trial Investigating the Efficacy and Safety of Visugromab and Nivolumab With or Without Docetaxel Versus Docetaxel in 2L Treatment of Participants With Metastatic NSCLC (GDFATHER-NSCLC-02)
Brief Title: Trial Investigating Visugromab and Nivolumab With or Without Docetaxel in 2L Treatment of Participants With Metastatic NSCLC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: CatalYm GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CTL-002-004; 2024-516794-70-00 (EU CTIS Number)
Record Dates: First submitted 2025-11-19; First posted 2025-11-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Metastatic Non-Squamous Non-Small Cell Lung Cancer; Adult Solid Tumor
Keywords: CTL-002; Visugromab; GDF-15
MeSH Terms: interventions — Nivolumab; Saline Solution; Docetaxel

STUDY DESIGN:
Intervention Model Description: Part A: Safety Run-In
  Part B and C: Randomized Part consists of 4 Arms:
  Arm A: Visugromab at the recommended dose for expansion (RDE) with Nivolumab and Docetaxel,
  Arm B: Visugromab 6 mg/kg with Nivolumab and Docetaxel,
  Arm C: Visugromab at the RDE with Nivolumab and Placebo (saline),
  Arm D: Double Placebo (saline) and Docetaxel
  Participants will be allocated in 2:1:1:1 ratio to treatment arms A, B, C, or D
Who Masked: Participant, Investigator
Masking Description: Throughout the randomized part of the trial, participants, Investigators, trial-assigned site staff (except for the pharmacists), the CRO (except for the unblinded clinical monitoring team), and imaging vendor will remain blinded to the information of which participant is receiving which IMP. Sponsor staff may be unblinded on an as needed basis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Arm A (Experimental): Visugromab (RDE) + Nivolumab (360 mg) + Docetaxel (75 mg/m2), intravenous (IV) on Day 1 of every 21-day cycle every 3 weeks (Q3W)
  Interventions: Biological: Visugromab RDE (recommended dose for expansion); Biological: Nivolumab; Drug: Docetaxel
- Arm B (Experimental): Visugromab (6mg/kg) + Nivolumab (360 mg) + Docetaxel (75 mg/m2), intravenous (IV) on Day 1 of every 21-day cycle every 3 weeks (Q3W)
  Interventions: Biological: Visugromab 6mg/kg; Biological: Nivolumab; Drug: Docetaxel
- Arm C (Experimental): Visugromab (RDE) + Nivolumab (360 mg) + Placebo (Saline) intravenous (IV) on Day 1 of every 21-day cycle every 3 weeks (Q3W)
  Interventions: Biological: Visugromab RDE (recommended dose for expansion); Biological: Nivolumab; Other: Placebo Saline Infusion
- Arm D (Active Comparator): Double Placebo (Saline) + Docetaxel (75 mg/m2), intravenous (IV) on Day 1 of every 21-day cycle (every 3 weeks, or Q3W)
  Interventions: Other: Placebo Saline Infusion; Drug: Docetaxel

INTERVENTIONS:
Biological: Visugromab RDE (recommended dose for expansion) — Participants receive Visugromab (RDE) intravenous (IV) on Day 1 of every 21-day cycle (every 3 weeks, or Q3W)
  Other Names: CTL-002
  Arms: Arm A; Arm C
Biological: Visugromab 6mg/kg — Participants receive Visugromab (6mg/kg) intravenous (IV) on Day 1 of every 21-day cycle (every 3 weeks, or Q3W)
  Other Names: CTL-002
  Arms: Arm B
Biological: Nivolumab — Participants receive Nivolumab 360mg intravenous (IV) on Day 1 of every 21-day cycle (every 3 weeks, or Q3W)
  Other Names: OPDIVO®
  Arms: Arm A; Arm B; Arm C
Other: Placebo Saline Infusion — Participants receive Saline intravenous (IV) on Day 1 of every 21-day cycle (every 3 weeks, or Q3W)
  Other Names: 0.9% NaCl
  Arms: Arm C; Arm D
Drug: Docetaxel — Participants receive Docetaxel 75 mg/m2 intravenous (IV) on Day 1 of every 21-day cycle (every 3 weeks, or Q3W)
  Arms: Arm A; Arm B; Arm D

SUMMARY:
This is an exploratory, signal-finding, randomized, placebo-controlled, blinded, multi-center phase 2b trial of the anti-GDF-15 antibody Visugromab (CTL-002) at two different dose levels plus Nivolumab with Docetaxel versus Visugromab at the higher dose plus Nivolumab with placebo versus double-placebo with Docetaxel, in participants that receive second-line treatment for non-squamous NSCLC after failure of prior first-line treatment including a CPI (checkpoint inhibitor).

The trial consists of 3 Parts: an open-label Safety Run-in part (Part A) followed by a subsequent randomized phase 2b part with 4 treatment arms. After the treatment of 15 participants with visugromab at the expansion dose, an interim safety and preliminary efficacy analysis will be conducted (Part B), followed by the treatment of the remaining participants (Part C).

ELIGIBILITY:
Main Inclusion Criteria:

* Participants must have histologically or cytologically confirmed diagnosis of stage IV non-squamous NSCLC.
* Participants must have demonstrated absence of actionable mutations (e.g. EGFR, ALK, among others) that suggest/require treatment with available targeted agent.
* Participants must have failed one line of prior systemic treatment for metastatic NSCLC containing an approved anti PD (L)1 checkpoint inhibitor (CPI). The minimum treatment duration on this regimen must have been 12 weeks exposure for the CPI with no documented progression in this period. Failure of the prior line of systemic treatment for metastatic NSCLC must have occurred under ongoing CPI treatment. Discontinuation of the prior CPI and line of treatment due to AEs, or any other reason than progression/relapse does not permit enrollment.
* Participants must have measurable disease determined by the local site Investigator by their assessment per RECIST v1.1.
* Participants must have life expectancy of at least 3 months as assessed by the Investigator.
* Participants must have ECOG performance status ≤1.

Main Exclusion Criteria:

* Participants must not have received more than one line of prior systemic treatment for advanced/metastatic NSCLC.
* Participants must not have a prior malignancy requiring treatment.
* Participants must not have a known or detected clinically active central nervous system (CNS) involvement by NSCLC or other tumors, e.g., with symptomatic metastases and/or carcinomatous meningitis
* Participants must not have any active autoimmune disease that has required systemic treatment in past 3 months before planned treatment start (i.e., with use of disease modifying agents, corticosteroids, or immunosuppressive drugs).
* Participants must not have interstitial lung disease or a history of (non-infectious) pneumonitis that required systemic steroids or current pneumonitis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 131 (Estimated)
Dates: Start 2025-10-07 (Actual); Primary Completion 2029-10-01 (Estimated); Study Completion 2031-10-01 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | up to 36 months
  Percentage of participants with a best overall response (BOR) of complete response (CR) or partial response (PR) per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 as assessed by the Investigator at any time during the core trial period

SECONDARY OUTCOMES:
Adverse Events | up to 60 months
  Incidence, type and severity of adverse events, treatment emergent adverse events, treatment-related adverse events and serious adverse events
CR rate | up to 36 months
  Complete response rate
PR rate | up to 36 months
  Partial response rate
ORR rate | up to 36 months
  Overall response rate
DOR | up to 36 months
  Duration of response
TTR | up to 36 months
  Time-to-respond
PFS | up to 60 months
  Progression-free survival
OS | up to 60 months
  Overall survival
Participant weight course over time | up to 39 months
  Participant weight course over time
Maximum Concentration (Cmax) of visugromab | up to 36 months
  Cmax is the maximum observed serum concentration of visugromab.
Minimum Concentration (Cmin) visugromab | up to 36 months
  Cmin is the minimum observed serum concentration of visugromab
Participants' subjective well-being as assessed by Non-Small Cell Lung Cancer Symptom Assessment Questionnaire (NSCLC-SAQ) | up to 39 months
  NSCLC-SAQ is a participant reported outcome with seven (7) items assessing five (5) symptom domains of NSCLC: cough, fatigue, pain, dyspnea, and appetite. Each item is scored individually from 0 ("None/Never") to 4 ("Severe/Always").
  The total score is calculated by summing domain scores, which are derived as follows: single-item domains (cough, dyspnea, appetite) use the item score; fatigue uses the mean of two items (or one if only one is answered); pain uses the highest score of two items (or one if only one is answered). The total score ranges from 0-20, with higher scores indicating more severe symptoms. If any domain score is missing, a total score is not computed

CONTACTS AND LOCATIONS:
Overall Officials: Lena Lemke, MD, Study Director — CatalYm GmbH
Locations (5):
- United States (2):
  - University of Alabama at Birmingham (O'Neal Comprehensive Cancer Center), Birmingham, Alabama
  - Duke University Medical Center, Durham, North Carolina
- University Hospital of Jaen, Jaén, Andalusia, Spain
- Switzerland (2):
  - University Hospital Basel, Basel
  - Cantonal Hospital Saint Gallen, Clinic of Oncology and Hematology, Sankt Gallen

IPD SHARING:
Plan to Share IPD: No